CLINICAL TRIAL: NCT03429335
Title: Just TRAC It! Transitioning Responsibly to Adult Care Using Smart Phone Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Just TRAC It!
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-02

CONDITIONS: Congenital Heart Disease; Heart; Surgery, Heart, Functional Disturbance as Result
Keywords: Transition; Adolescents; Smart phone
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Patients will be randomized individually in permuted blocks with randomly varying sizes of 2 and 4, and allocation ratio 1:1 for intervention and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teaching session & Just TRAC It (Experimental): Youth will attend a single one-on-one teaching session with a cardiology nurse (RN) the same day as their pediatric cardiology clinic visit. The RN will also explain "Just TRAC It!" and help the youth to enter their health information into their phone.
  Interventions: Behavioral: Teaching session; Behavioral: Just TRAC It!
- Teaching session & MyHealth Passport (Active Comparator): Youth will attend a single one-on-one teaching session with a cardiology nurse (RN) the same day as their pediatric cardiology clinic visit. The RN will help youth complete and print out a "MyHealth Passport" to track their medical information.
  Interventions: Behavioral: Teaching session; Behavioral: MyHealth Passport

INTERVENTIONS:
Behavioral: Teaching session — The cardiology nurse (RN) will have an hour long one-on-one teaching session prior to their pediatric cardiology clinic visit. The RN will go over the youth's cardiac history including the chronic heart disease diagnoses, names and dates of cardiac surgical procedures and cardiac catheterizations, and current cardiac medications and doses. She will also discuss transitioning from pediatric to adult care and healthy lifestyle choices.
Behavioral: Just TRAC It! — Just TRAC It! (Transitioning Responsibly to Adult Care) is a mobile health intervention that encourages youth to use existing functions on their personal phones to track their health information. The use of Just TRAC It! allows youth to electronically document all medical information that would previously be printed on their MyHealth Passport, but may offer additional functionality in terms of learning to manage their health.
  Arms: Teaching session & Just TRAC It
Behavioral: MyHealth Passport — MyHealth Passport is a customized, wallet-size card that includes the youth's important medical information. The RN will help the youth create a MyHealth Passport online, and print out the card for them.
  The same educational intervention will be completed by cardiology nurse using a MyHealth Passport to track their medical information instead of the electronic "Just TRAC It!"
  Arms: Teaching session & MyHealth Passport

SUMMARY:
The Just TRAC It! study (Transitioning Responsibly to Adult Care using smart phone technology) is a randomized controlled trial designed to evaluate the impact of using smart phone technology in combination with the nurse led transition intervention, versus the current standard of care (nurse led transition intervention including MyHealth Passport), on preparing adolescents with chronic cardiac disease to successfully transition from pediatric to adult cardiology care. "Just TRAC it!" is a mobile-health intervention designed to teach youth to manage their health using existing functions on their mobile devices. We propose to conduct a nurse-led intervention that encourages adolescents to use "Just TRAC it!" while addressing the healthcare transition needs of 16-18 year olds.

DETAILED DESCRIPTION:
Many adolescents and young adults living with chronic health conditions lack knowledge about their medical condition and confidence communicating with health care providers. Despite various positions statements on transition by the Canadian Pediatric Society, the American Academy of Pediatrics and the American Heart Association, there is limited evidence on the impact and effectiveness of transition interventions. Due to the convenience and accessibility of technology, adolescents embrace technology-based interventions to aid in their disease management and to improve their transition experience. However, there is a paucity of evidence-based apps in contrast to countless existing apps that are not evidence-based, which act as a barrier to physicians prescribing them. There is a pressing need for credible evidence on the effectiveness and value of health apps in improving self-management skills in adolescents.

Instead of redesigning a mobile app, the Just TRAC It! encourages youth to use existing functions on their personal phones to track their health information. This information is easily retrievable when visiting health care providers and can help youth take ownership in managing their own health. This free option, using the technology already on most phones, can be used for any patient population or disease category. The use of Just TRAC It! allows youth to electronically document all medical information that would previously be printed on their MyHealth Passport, but may offer additional functionality in terms of learning to manage their health. Further investigation is warranted to evaluate the effectiveness of Just TRAC It! on improving patient knowledge, self-management skills, and transition readiness.

The Stollery Children's Hospital is an international leader in pediatric to adult cardiology transition research, with two randomized clinical trials completed (CHAPTER 1 Trial, Mackie et al, Heart 2014 and CHAPTER 2 Trial, Mackie et al, BMC Cardiovascular 2016) and a 3rd in progress. The Just Trac It! Trial is an extension of our prior work. The results of the CHAPTER 1 Trial inform the current standard of care for transition interventions currently offered to all 16-18 year olds in our program who have had prior cardiac surgery, and this standard of care is the "usual care" (control) group for the Just Trac It! Study.

ELIGIBILITY:
Inclusion Criteria:

* 16-18 year olds with moderate or complex CHD, or acquired heart disease requiring surgery (e.g., rheumatic heart disease, prior endocarditis, prior valve replacement, Marfan's syndrome) who are followed at the Stollery Children's Hospital.

Exclusion Criteria:

* less than grade 6 level of reading and comprehension based on parent report
* heart transplantation, as this results in distinct health challenges
* does not have a personal mobile device, as this is required for the Just TRAC It! intervention

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in transition readiness measured by the TRANSITION-Q Questionnaire score | 3 months
  This 14-item instrument, developed at McMaster University, is written at a grade 4.4 level and takes about 3 minutes to complete.
Change in transition readiness measured by the TRANSITION-Q Questionnaire score | 6 months
  This 14-item instrument, developed at McMaster University, is written at a grade 4.4 level and takes about 3 minutes to complete.

SECONDARY OUTCOMES:
Frequency of use and perceived helpfulness of intervention measured by Just TRAC It! Questionnaire | 3 months
  This questionnaire was developed for the purpose of this study to ascertain perceived helpfulness and frequency of use.
Frequency of use and perceived helpfulness of intervention measured by Just TRAC It! Questionnaire | 6 months
  This questionnaire was developed for the purpose of this study to ascertain perceived helpfulness and frequency of use.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Mackie, MD, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campbell F, Biggs K, Aldiss SK, O'Neill PM, Clowes M, McDonagh J, While A, Gibson F. Transition of care for adolescents from paediatric services to adult health services. Cochrane Database Syst Rev. 2016 Apr 29;4(4):CD009794. doi: 10.1002/14651858.CD009794.pub2. PMID 27128768
- [Background] Van Deyk K, Pelgrims E, Troost E, Goossens E, Budts W, Gewillig M, Moons P. Adolescents' understanding of their congenital heart disease on transfer to adult-focused care. Am J Cardiol. 2010 Dec 15;106(12):1803-7. doi: 10.1016/j.amjcard.2010.08.020. Epub 2010 Nov 2. PMID 21126624
- [Background] Kantoch MJ, Collins-Nakai RL, Medwid S, Ungstad E, Taylor DA. Adult patients' knowledge about their congenital heart disease. Can J Cardiol. 1997 Jul;13(7):641-5. PMID 9251576
- [Background] Dore A, de Guise P, Mercier LA. Transition of care to adult congenital heart centres: what do patients know about their heart condition? Can J Cardiol. 2002 Feb;18(2):141-6. PMID 11875583
- [Background] Clarizia NA, Chahal N, Manlhiot C, Kilburn J, Redington AN, McCrindle BW. Transition to adult health care for adolescents and young adults with congenital heart disease: perspectives of the patient, parent and health care provider. Can J Cardiol. 2009 Sep;25(9):e317-22. doi: 10.1016/s0828-282x(09)70145-x. PMID 19746251
- [Background] Moons P, Pinxten S, Dedroog D, Van Deyk K, Gewillig M, Hilderson D, Budts W. Expectations and experiences of adolescents with congenital heart disease on being transferred from pediatric cardiology to an adult congenital heart disease program. J Adolesc Health. 2009 Apr;44(4):316-22. doi: 10.1016/j.jadohealth.2008.11.007. Epub 2009 Feb 12. PMID 19306789
- [Background] Transition to adult care for youth with special health care needs. Paediatr Child Health. 2007 Nov;12(9):785-93. doi: 10.1093/pch/12.9.785. No abstract available. PMID 19030468
- [Background] American Academy of Pediatrics; American Academy of Family Physicians; American College of Physicians-American Society of Internal Medicine. A consensus statement on health care transitions for young adults with special health care needs. Pediatrics. 2002 Dec;110(6 Pt 2):1304-6. PMID 12456949
- [Background] Sable C, Foster E, Uzark K, Bjornsen K, Canobbio MM, Connolly HM, Graham TP, Gurvitz MZ, Kovacs A, Meadows AK, Reid GJ, Reiss JG, Rosenbaum KN, Sagerman PJ, Saidi A, Schonberg R, Shah S, Tong E, Williams RG; American Heart Association Congenital Heart Defects Committee of the Council on Cardiovascular Disease in the Young, Council on Cardiovascular Nursing, Council on Clinical Cardiology, and Council on Peripheral Vascular Disease. Best practices in managing transition to adulthood for adolescents with congenital heart disease: the transition process and medical and psychosocial issues: a scientific statement from the American Heart Association. Circulation. 2011 Apr 5;123(13):1454-85. doi: 10.1161/CIR.0b013e3182107c56. Epub 2011 Feb 28. No abstract available. PMID 21357825
- [Background] Mackie AS, Islam S, Magill-Evans J, Rankin KN, Robert C, Schuh M, Nicholas D, Vonder Muhll I, McCrindle BW, Yasui Y, Rempel GR. Healthcare transition for youth with heart disease: a clinical trial. Heart. 2014 Jul;100(14):1113-8. doi: 10.1136/heartjnl-2014-305748. Epub 2014 May 19. PMID 24842870
- [Background] Huang JS, Gottschalk M, Pian M, Dillon L, Barajas D, Bartholomew LK. Transition to adult care: systematic assessment of adolescents with chronic illnesses and their medical teams. J Pediatr. 2011 Dec;159(6):994-8.e2. doi: 10.1016/j.jpeds.2011.05.038. Epub 2011 Jul 23. PMID 21784450
- [Background] Trawley S, Browne JL, Hagger VL, Hendrieckx C, Holmes-Truscott E, Pouwer F, Skinner TC, Speight J. The Use of Mobile Applications Among Adolescents with Type 1 Diabetes: Results from Diabetes MILES Youth-Australia. Diabetes Technol Ther. 2016 Dec;18(12):813-819. doi: 10.1089/dia.2016.0233. Epub 2016 Oct 27. PMID 27788032
- [Background] Geryk LL, Roberts CA, Sage AJ, Coyne-Beasley T, Sleath BL, Carpenter DM. Parent and Clinician Preferences for an Asthma App to Promote Adolescent Self-Management: A Formative Study. JMIR Res Protoc. 2016 Dec 6;5(4):e229. doi: 10.2196/resprot.5932. PMID 27923777
- [Background] Crosby LE, Ware RE, Goldstein A, Walton A, Joffe NE, Vogel C, Britto MT. Development and evaluation of iManage: A self-management app co-designed by adolescents with sickle cell disease. Pediatr Blood Cancer. 2017 Jan;64(1):139-145. doi: 10.1002/pbc.26177. Epub 2016 Aug 30. PMID 27574031
- [Background] Majeed-Ariss R, Baildam E, Campbell M, Chieng A, Fallon D, Hall A, McDonagh JE, Stones SR, Thomson W, Swallow V. Apps and Adolescents: A Systematic Review of Adolescents' Use of Mobile Phone and Tablet Apps That Support Personal Management of Their Chronic or Long-Term Physical Conditions. J Med Internet Res. 2015 Dec 23;17(12):e287. doi: 10.2196/jmir.5043. PMID 26701961
- [Background] Misra S, Lewis TL, Aungst TD. Medical application use and the need for further research and assessment for clinical practice: creation and integration of standards for best practice to alleviate poor application design. JAMA Dermatol. 2013 Jun;149(6):661-2. doi: 10.1001/jamadermatol.2013.606. No abstract available. PMID 23783150
- [Background] Huang JS, Terrones L, Tompane T, Dillon L, Pian M, Gottschalk M, Norman GJ, Bartholomew LK. Preparing adolescents with chronic disease for transition to adult care: a technology program. Pediatrics. 2014 Jun;133(6):e1639-46. doi: 10.1542/peds.2013-2830. Epub 2014 May 19. PMID 24843066
- [Background] Klassen AF, Grant C, Barr R, Brill H, Kraus de Camargo O, Ronen GM, Samaan MC, Mondal T, Cano SJ, Schlatman A, Tsangaris E, Athale U, Wickert N, Gorter JW. Development and validation of a generic scale for use in transition programmes to measure self-management skills in adolescents with chronic health conditions: the TRANSITION-Q. Child Care Health Dev. 2015 Jul;41(4):547-58. doi: 10.1111/cch.12207. Epub 2014 Oct 28. PMID 25351414
- [Background] Boutron I, Moher D, Altman DG, Schulz KF, Ravaud P; CONSORT Group. Methods and processes of the CONSORT Group: example of an extension for trials assessing nonpharmacologic treatments. Ann Intern Med. 2008 Feb 19;148(4):W60-6. doi: 10.7326/0003-4819-148-4-200802190-00008-w1. PMID 18283201